CLINICAL TRIAL: NCT05174195
Title: Can a Three Months Treatment With Oral Desogestrel Prior to Insertion of the Etonogestrel Subdermal Implant Improve Continuation Rate at One Year?
Brief Title: Does Oral Desogestrel Prior to Insertion of the Etonogestrel Subdermal Implant Improve Continuation Rate at One Year?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult recruitment
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Michal Yaron, Head of Unit Ambulatory Gynecology, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCER 16-972
Record Dates: First submitted 2021-07-29; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Contraception; Progestogen Adverse Reaction

STUDY DESIGN:
Intervention Model Description: Randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESI (Implanon NXT® subdermal implant) (Active Comparator): In this group, the implant was inserted immediately after thorough explanations of the potential side effects and possible adverse events
  Interventions: Drug: Implanon NXT® subdermal implant
- DSG + ESI(Desogestrel +Implanon NXT® subdermal implant) (Experimental): In this group, patients were given a 3 months' supply of 75µg of DSG to be started immediately after which insertion of an ESI was proposed. Similarly, explanations of the potential side effects and possible adverse events were presented to the patient before treatment initiation.
  Interventions: Drug: Desogestrel 0.075 milligram; Drug: Implanon NXT® subdermal implant

INTERVENTIONS:
Drug: Desogestrel 0.075 milligram — Inserted after 3 months use of DESOGESTREL
  Other Names: Implanon NXT® subdermal implant
  Arms: DSG + ESI(Desogestrel +Implanon NXT® subdermal implant)
Drug: Implanon NXT® subdermal implant — Inserted immediately

SUMMARY:
Objective: The etonogestrel subdermal implant (ESI) is an effective and safe method of contraception. Although highly efficient, ESI produces often side effects that reduce its tolerance and acceptance. Daily oral desogestrel (DSG) prior to the insertion of ESI might help reduce its premature discontinuation. Our aim was to evaluate if this pre-treatment increases ESI's tolerance.

Methods: Between 15.08.2016 and 30.09.2019, the investigators conducted a randomized prospective study of women aged 18 to 42 years who were interested to use Implanon and were willing to have 90 days of pre-treatment with DSG, in the family planning clinic of the Geneva University Hospitals and the Hospital of Basel. Women were randomized into either the study ESI only group or to the DSG + ESI group. In the DSG + ESI group, patients were given a 3 months' supply of 75µg of DSG before the insertion of the ESI.

A 3 months visit was pre-programmed for all participants where the bleeding calendar and the questionnaires were collected. All patients were called over the phone after 12 months post ESI insertion in both groups.

DETAILED DESCRIPTION:
Study and treatment periods

1 year of patient recruitment 15 months of follow up (90 days OD plus 1 year Implant or 1 year Implant)

Measurements and Procedures:

Assessment of premature ablation (PA) in months 3-12 (ESI only) or 3-15 (OD+ESI). This will require a contact with all patients at 12/15 months to verify if implant is still in place, and if it was removed, why (and possibly to also reassess symptoms).

Women with known PA can be exempted from this follow-up. In case of PA, reasons will be explored and questioned.

* Assessment of symptoms at 3 months only (bleeding calendar and satisfaction questionnaire, see below)
* Assessment of willingness to receive implant at 3 months in OD+ESI group data collection is limited to these items, in order to limit burden on participants, and to focus resources on high quality of data (as opposed to quantity).

ELIGIBILITY:
Inclusion criteria:

* Women age of 18 - 42 years
* Interested in the use of ESI
* Accepting to have 90 days pre-treatment with OD
* Signed informed consent

Exclusion criteria:

* Pregnancy
* Lactation,
* vaginal bleeding of unknown origin,
* wish to become pregnant,
* weight over 80 kg,
* history of deep vein thrombosis/Pulmanory embolism,
* hypertension,
* Diabetes or other metabolic diseases,
* coagulation disorders,
* severe hepatic disorder,
* history of breast/endometrial cancer,
* known hypersensitivity to study drug,
* current treatment with enzyme inducing drugs (e.g.: phenytoin, carbamazepine, phenobarbital, etc.)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Tolerance of Implanon | at 1 year after implant insertion (or at ablation)
  self-reported

SECONDARY OUTCOMES:
Discontinuation of implant, | at any time after insertion through study completion, an average of 1 year
  frequency of ablation of any cause and due to intolerance
  * severity of specific symptoms at 1 year (or at ablation)
  * severity of specific symptoms at 1 year (or at ablation)
specific symptoms | at 1 year after implant insertion
  measured by questionnaires on bleeding patterns and satisfaction on a Likert scale

REFERENCES:
- [Derived] Lombardi Fah V, Catarino R, Castillo S, Badda M, Gezer-Dickschat S, Thieringer F, Tschudin S, Viviano M, Yaron M. Can a 3 months treatment with oral Desogestrel prior to insertion of the etonogestrel-releasing contraceptive implant improve continuation rate at 1 year? A randomized trial. BMC Res Notes. 2023 Mar 13;16(1):35. doi: 10.1186/s13104-023-06304-3. PMID 36915205